CLINICAL TRIAL: NCT01611974
Title: A Phase 2, Randomized Study to Assess the Safety and Anti-cytomegalovirus (CMV) Activity of Different Doses of Maribavir for Treatment of CMV Infections That Are Resistant or Refractory to Treatment With Ganciclovir/Valganciclovir or Foscarnet in Transplant Recipients
Brief Title: Maribavir for Treatment of Resistant or Refractory CMV Infections in Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1263-202; SHP620-202 (Other: Shire Development LLC)
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Cytomegalovirus (CMV)
Keywords: transplant; treatment; resistant; CMV; refractory; cytomegalovirus
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Maribavir 400 mg twice daily (Experimental)
  Interventions: Drug: Maribavir
- Maribavir 800 mg twice daily (Experimental)
  Interventions: Drug: Maribavir
- Maribavir 1200 mg twice daily (Experimental)
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Tablet for oral administration

SUMMARY:
This study will assess safety, antiviral activity, and pharmacokinetics of different doses of maribavir administered orally for up to 24 weeks for treatment of CMV infections that are resistant or refractory to treatment with ganciclovir/valganciclovir or foscarnet in recipients of stem cell or solid organ transplants.

ELIGIBILITY:
Inclusion Criteria

1. Be ≥12 years of age.
2. Weigh ≥ 40 kg.
3. Be a recipient of stem cell or solid organ transplantation.
4. Have documented CMV infection in blood or plasma, with a screening value of ≥1,000 DNA copies/mL.
5. Have a current CMV infection that is resistant (known CMV genetic mutations) or refractory (clinical failure to respond) to treatment with ganciclovir/valganciclovir and/or foscarnet.
6. If female, be either postmenopausal, surgically sterile, or have a negative pregnancy test prior to randomization.
7. Be able to swallow tablets.
8. If adult, provide written informed consent. If child (age <18 years), have a parent/legal guardian who is willing and able to provide written informed consent (with assent from the child when appropriate).
9. Be assessed by the investigator to determine whether prophylaxis for non-CMV herpesvirus infections (e.g., herpes simplex virus [HSV type 1 and type 2] and varicella zoster virus [VZV]) is appropriate according to institutional guidelines or standard practices, keeping in mind that maribavir is not active in vitro against these viruses.

Exclusion Criteria

1. Be receiving any other anti-CMV agent(s).
2. Have a current CMV infection that is considered resistant or refractory due to inadequate adherence to prior oral anti-CMV treatment.
3. Have severe vomiting, diarrhea, or other severe gastrointestinal illness within 24 hours prior to the time of enrollment.
4. Have severe hepatic impairment.
5. Require mechanical ventilation or vasopressors for hemodynamic support at the time of enrollment.
6. Have expected survival less than 6 weeks.
7. Be pregnant or breastfeeding.
8. Other clinically significant medical or surgical condition.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2014-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (32):
- United States (32):
  - UCLA Medical Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health Care System, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Methodist Healthcare System, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Sun K, Fournier M, Sundberg AK, Song IH. Maribavir: Mechanism of action, clinical, and translational science. Clin Transl Sci. 2024 Jan;17(1):e13696. doi: 10.1111/cts.13696. PMID 38071422
- [Derived] Chou S, Song K, Wu J, Bo T, Crumpacker C. Drug Resistance Mutations and Associated Phenotypes Detected in Clinical Trials of Maribavir for Treatment of Cytomegalovirus Infection. J Infect Dis. 2022 Sep 4;226(4):576-584. doi: 10.1093/infdis/jiaa462. PMID 32726419
- [Derived] Papanicolaou GA, Silveira FP, Langston AA, Pereira MR, Avery RK, Uknis M, Wijatyk A, Wu J, Boeckh M, Marty FM, Villano S. Maribavir for Refractory or Resistant Cytomegalovirus Infections in Hematopoietic-cell or Solid-organ Transplant Recipients: A Randomized, Dose-ranging, Double-blind, Phase 2 Study. Clin Infect Dis. 2019 Apr 8;68(8):1255-1264. doi: 10.1093/cid/ciy706. PMID 30329038
- [Derived] Schubert A, Ehlert K, Schuler-Luettmann S, Gentner E, Mertens T, Michel D. Fast selection of maribavir resistant cytomegalovirus in a bone marrow transplant recipient. BMC Infect Dis. 2013 Jul 19;13:330. doi: 10.1186/1471-2334-13-330. PMID 23870704

RESULTS

PARTICIPANT FLOW:
Groups:
- Maribavir 400 mg Twice Daily: Participants received oral maribavir at 400 mg twice daily for a maximum duration of 24 weeks. Participants were then followed for 12 weeks.
- Maribavir 800 mg Twice Daily: Participants received oral maribavir at 800 mg twice daily for a maximum duration of 24 weeks. Participants were then followed for 12 weeks.
- Maribavir 1200 mg Twice Daily: Participants received oral maribavir at 1200 mg twice daily for a maximum duration of 24 weeks. Participants were then followed for 12 weeks.
Period: Overall Study
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Started | 40 | 40 | 40
Completed | 25 | 25 | 24
Not Completed | 15 | 15 | 16
Not completed — Death | 10 | 12 | 10
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 5 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat Safety population, defined as all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (14.25) | 55.4 (14.13) | 50.0 (12.96) | 52.5 (13.86)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 11 | 10 | 14 | 35
  45 to 64 years | 22 | 18 | 20 | 60
  65 to 75 years | 7 | 12 | 6 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 16 | 51
  Male | 21 | 24 | 24 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Undetectable Plasma Cytomegalovirus (CMV) Within 6 Weeks
Description: Blood samples were collected at the study sites, processed to plasma aliquots, and sent to the central laboratory for quantitative CMV DNA polymerase chain reaction (PCR) testing. Plasma samples were assayed for CMV concentration using a qualified PCR method. This method was linear over 200-100,000 viral copies/mL with a lower limit of quantification (LLOQ) of 200 copies/mL. Results below LLOQ were considered undetectable. Confirmed undetectable plasma CMV DNA within 6 weeks was defined as 2 consecutive post-baseline, on-treatment undetectable results separated by >/= 5 days (assessed by the central laboratory). Samples were collected on Days 1 and 8, weekly during Weeks 2-6, and once in Weeks 8, 10, 12, 16, 20, 24 (treatment) and Weeks 1, 4, 8, 12 (follow-up). Permissible assessment windows were: Days 8-15 +/- 1 day; Weeks 3-4 +/- 2 days; Weeks 5-6 +/- 3 days; Weeks 8-12 +/- 4 days; Weeks 16-24 +/- 7 days (treatment) and Weeks 1-4 +/- 2 days; Weeks 8-12 +/- 4 days (follow-up).
Time Frame: 6 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 40 | 40 | 38
participants | 28 | 25 | 27

2. Primary Outcome: Number of Participants With a Treatment Emergent Adverse Event (TEAE).
Description: Treatment-emergent adverse events are those events that occurred on or after study drug administration through 7 days after the last dose of study drug, or are events that occurred prior to study drug administration and recurred with increased severity after taking study drug through 7 days after the last dose of study drug.
Time Frame: 25 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 40 | 40 | 40
participants
  Any TEAE | 40 | 40 | 40
  Serious TEAE | 28 | 27 | 26

3. Secondary Outcome: Number of Participants With CMV Recurrence
Description: Blood samples were collected at the study sites, processed to plasma aliquots, and sent to the central laboratory for quantitative CMV DNA polymerase chain reaction (PCR) testing. Plasma samples were assayed for CMV concentration using a qualified PCR method. CMV recurrence was defined as achievement of undetectable plasma CMV DNA at any time after Day 1 in at least 2 consecutive samples separated by at least 5 days, followed by detectable plasma CMV DNA in at least 2 consecutive samples separated by at least 5 days (assessed by the central laboratory). For the analyses of CMV recurrence, the first of 2 consecutive confirmed undetectable plasma CMV DNA results had to be on-treatment. CMV DNA PCR values of ≥200 copies/mL were considered detectable. Participants assessed for recurrence (n= 29, 27, 30) are the subset of the ITT-S who had at least 2 consecutive undetectable plasma CMV DNA results separated by at least 5 days, including early withdrawn qualified subjects.
Time Frame: 36 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 40 | 40 | 40
participants | 7 | 11 | 12

4. Secondary Outcome: Time to First Confirmed Undetectable Plasma CMV DNA Within 6 Weeks and at Any Time During The Study
Description: Blood samples were collected at the study sites, processed to plasma aliquots, and sent to the central laboratory for quantitative CMV DNA polymerase chain reaction (PCR) testing. Plasma samples were assayed for CMV concentration using a qualified PCR method. The time to event was defined as the time from first dose of study drug to first undetectable plasma CMV DNA within 6 weeks and at any time during the study, defined as the date of the first of at least 2 consecutive post-baseline, on-treatment undetectable results (<200 copies/mL) separated by at least 5 days; as assessed by the central laboratory. The median values are Kaplan-Meier estimates.
Time Frame: 6 weeks after start of treatment, within 36 weeks of start of treatment
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 40 | 40 | 40
days
  Within 6 weeks, n = 40, 40, 38 | 24.0 [15.0 to 31.0] | 28.0 [15.0 to 36.0] | 22.0 [15.0 to 28.0]
  Anytime during the study, n = 40, 40, 40 | 24.0 [15.0 to 31.0] | 28.0 [15.0 to 38.0] | 22.0 [19.0 to 30.0]

5. Secondary Outcome: Time to CMV Recurrence
Description: Blood samples were collected at the study sites, processed to plasma aliquots, and sent to the central laboratory for quantitative CMV DNA polymerase chain reaction (PCR) testing. Plasma samples were assayed for CMV concentration using a qualified PCR method. The time to event was defined as the time of the first of at least 2 consecutive samples, separated by at least 5 days, with detectable plasma CMV DNA after achievement of undetectable plasma CMV DNA in at least 2 consecutive samples, separated by at least 5 days, at any time after Day 1; as assessed by the central laboratory. Participants assessed for recurrence (n= 29, 27, 30) are the subset of the ITT-S who had at least 2 consecutive undetectable plasma CMV DNA results separated by at least 5 days, including early withdrawn qualified subjects. The median values are Kaplan-Meier estimates.
Time Frame: 36 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 40 | 40 | 40
days | NA [NA to NA] — The median and 95% CIs were not estimable. | 118.0 [37.0 to NA] — The upper 95% CI was not estimable. | 161.0 [92.0 to NA] — The upper 95% CI was not estimable.

6. Secondary Outcome: Maximum Concentration (Cmax) of Maribavir
Description: For the subset of participants who had pharmacokinetic (PK) profiling performed, non-compartmental PK analyses were used to determine Cmax, time to Cmax (tmax), time of last non-zero concentration (tlast), area under the plasma concentration versus time curve from the time of dosing to the last measurable concentration (AUClast), and half-life (t½). Values below the LLOQ post-baseline were replaced with a value of 0 ug/mL. Values below the LLOQ at baseline were replaced with zero as it was assumed that subjects had no levels of maribavir at baseline. At the designated timepoints, the PK sample was obtained 2-4 hours after the dose of study drug; for subjects who were inpatients, a pre-dose PK sample also was collected. These samples were not required at Day 8 and Week 4 for subjects who had PK profiles performed on those days.
Time Frame: pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Day 8 and the Week 4 visit
Population: The Pharmacokinetic Profile Population, defined as all participants in the ITT-S Population who had plasma samples drawn and tested for maribavir concentrations
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 12 | 13 | 8
ug/mL
  Visit 3, n = 12, 10, 8 | 18.5 (7.39) | 35.1 (12.0) | 45.1 (21.2)
  Visit 6, n = 8, 10, 6 | 17.8 (8.36) | 25.0 (9.69) | 35.6 (25.8)

7. Secondary Outcome: Time to Maximum Concentration (Tmax) of Maribavir
Description: as for outcome 6
Time Frame: pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Day 8 and the Week 4 visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 12 | 13 | 8
hours
  Visit 3, n = 12, 10, 8 | 3.56 (2.99) | 2.70 (2.89) | 2.81 (2.02)
  Visit 6, n = 8, 10, 6 | 1.66 (0.765) | 3.23 (2.28) | 3.12 (1.05)

8. Secondary Outcome: Time of Last Non-Zero Concentration (Tlast) of Maribavir
Description: as for outcome 6
Time Frame: pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Day 8 and the Week 4 visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 12 | 13 | 8
hours
  Visit 3, n = 12, 10, 8 | 9.03 (2.55) | 8.26 (2.48) | 8.71 (1.45)
  Visit 6, n = 8, 10, 6 | 7.37 (3.70) | 7.99 (1.65) | 8.61 (1.64)

9. Secondary Outcome: Area Under The Plasma Concentration Versus Time Curve From The Time of Dosing to The Last Measurable Concentration (AUClast) of Maribavir
Description: as for outcome 6
Time Frame: pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Day 8 and the Week 4 visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 12 | 13 | 8
h*ug/mL
  Visit 3, n = 12, 10, 8 | 100 (50.4) | 179 (69.6) | 264 (147)
  Visit 6, n = 8, 10, 6 | 90.9 (64.3) | 139 (61.3) | 207 (161)

10. Secondary Outcome: Half-Life (T½) of Maribavir
Description: as for outcome 6
Time Frame: pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Day 8 and the Week 4 visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Number analyzed (Participants) | 12 | 13 | 8
hours
  Visit 3, n = 6, 7, 3 | 5.56 (3.85) | 6.08 (3.51) | 7.77 (3.59)
  Visit 6, n = 5, 5, 3 | 4.32 (1.25) | 6.34 (1.41) | 5.33 (2.55)

ADVERSE EVENTS:
Description: Treatment emergent AEs are reported for the Intent-to-Treat Safety Population, defined as all randomized participants who received at least 1 dose of study drug.
Arm/Group | Maribavir 400 mg Twice Daily | Maribavir 800 mg Twice Daily | Maribavir 1200 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 28/40 | 27/40 | 26/40
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maribavir 400 mg Twice Daily (N=40) | Maribavir 800 mg Twice Daily (N=40) | Maribavir 1200 mg Twice Daily (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 2 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 1 | 0 | 1
Lung transplant rejection (Immune system disorders) | 2 | 1 | 1
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0 | 1
Cytomegalovirus gastroenteritis (Infections and infestations) | 2 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 5 | 6
Encephalitis viral (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 1
Sepsis (Infections and infestations) | 2 | 3 | 1
Blood stem cell transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 2 | 3 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1 | 0
Encephalitis cytomegalovirus (Infections and infestations) | 0 | 1 | 0
Herpes simplex meningoencephalitis (Infections and infestations) | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Jejunal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Immunosuppresant drug level increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maribavir 400 mg Twice Daily (N=40) | Maribavir 800 mg Twice Daily (N=40) | Maribavir 1200 mg Twice Daily (N=40)
Dysgeusia (Nervous system disorders) | 24 | 25 | 29
Nausea (Gastrointestinal disorders) | 14 | 9 | 12
Vomiting (Gastrointestinal disorders) | 11 | 12 | 11
Cytomegalovirus infection (Infections and infestations) | 3 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 11 | 10
Fatigue (General disorders) | 7 | 10 | 7
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 10
Oedema peripheral (General disorders) | 11 | 5 | 6
Headache (Nervous system disorders) | 9 | 4 | 6
Renal impairment (Renal and urinary disorders) | 1 | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 7 | 6 | 3
Constipation (Gastrointestinal disorders) | 5 | 5 | 5
Pneumonia (Infections and infestations) | 5 | 3 | 4
Pyrexia (General disorders) | 4 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 4 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 5
Immunosuppressant drug level increased (Investigations) | 4 | 2 | 5
Urinary tract infection (Infections and infestations) | 6 | 2 | 2
Depression (Psychiatric disorders) | 2 | 8 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5
Hypotension (Vascular disorders) | 4 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 3
Clostridium difficile infection (Infections and infestations) | 2 | 2 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 4
Acute graft versus host disease (Immune system disorders) | 1 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 5 | 3
Weight decreased (Investigations) | 2 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
Ascites (Gastrointestinal disorders) | 3 | 1 | 3
Chills (General disorders) | 2 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1 | 3
Bacterial test positive (Investigations) | 2 | 3 | 1
Blood creatinine increased (Investigations) | 1 | 3 | 2
Fluid overload (Metabolism and nutrition disorders) | 4 | 1 | 0
Hepatic enzyme increased (Investigations) | 3 | 3 | 0
Hypertension (Vascular disorders) | 3 | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 1
Lung transplant rejection (Immune system disorders) | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 4 | 1
BK virus infection (Infections and infestations) | 3 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3
Local swelling (General disorders) | 2 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Pain (General disorders) | 2 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 3 | 1
Asthenia (General disorders) | 1 | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Generalised oedema (General disorders) | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 3 | 1
Malaise (General disorders) | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 2
Gait disturbance (General disorders) | 1 | 2 | 0
Genital herpes (Infections and infestations) | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 2 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 3
Visual impairment (Eye disorders) | 0 | 0 | 3
Weight increased (Investigations) | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 2
Libido decreased (Psychiatric disorders) | 0 | 0 | 2
Neutrophil count increased (Investigations) | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Swelling (General disorders) | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.